CLINICAL TRIAL: NCT00166907
Title: Balance Recovery and Training on Fall Prevention in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9100005692
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-06

CONDITIONS: Stroke
Keywords: Stroke; Balance; Proactive control; Reactive control; Recovery; Training; Fall
MeSH Terms: conditions — Stroke | interventions — Exercise

INTERVENTIONS:
Behavioral: Balance and Exercise

SUMMARY:
The specific aims of this research are delineated as the following: Aim 1: To investigate the neuromuscular and biomechanical mechanisms of the emerging processes of proactive and reactive balance control during sitting and standing in patients with stroke at different stages of the recovery course. Aim 2: To determine the relationships between brain lesion sites and the recovery patterns of reactive and proactive balance control mechanisms in patients with stroke. Aim 3: To determine the relationships between the impairments in reactive and proactive balance control mechanisms and functional outcome as well as fall incidence in patients following stroke. Aim 4: To investigate the efficacy of different training regimens in improving reactive and proactive balance control strategies and in preventing falls in stroke patients with different brain lesion sites. Principally, three hypotheses are to be tested: Hypothesis 1:The emerging processes and recovery patternes of proactive and reactive balance control may be different among stroke patients with different brain lesion locations. Hypothesis 2:There are positive correlations between the level of impairments in reactive and proactive balance control mechanisms and functional outcome as well as fall incidence in patients following stroke. Hypothesis 3:Training regimens that could best facilitate the emergence or improvement in reactive and proactive balance control strategies are different.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of chronic disability in the world. Falls are one of the primary complications after stroke. The incidence of falls ranges from 25% to 75% among stroke patients residing in different settings, with greater incidence of falls occurring after discharge home. Postural instability has been suggested as one of the main causes leading to falls in this population. The recovery of the ability to maintain balance during activities of daily living, therefore, is essential for functional independence and safety of these patients. In the following paragraphs, the knowledge gaps taht we are proposing to bridge in this study and the revelant literature that leads us to identify these gaps are discussed.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults

* between 45 and 75 years old
* having no neuromuscular or musculoskeletal disorders that would jeopardize their balance control abilities
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital

Stroke patients

* between 45 and 75 years old
* hemiplegic or hemiparetic as a result of a single cerebral vascular accident with brain lesions primarily involving one of the following areas: the primary motor cortex, supplementary motor/premotor areas, parietal cortex, or basal ganglia
* medically stable with no ongoing complications
* within 30 days post stroke able to independently sit without using any assistive device for at least 3 minutes if being tested on the 14th and 30th days post-stroke and able to stand and take a fast step independently in standing without using any assistive device for at least 3 minutes when tested on the 60th, 90th, 180th, 360th, 540th, and 720th days post stroke onset
* able to communicate with the experimenters
* having no hemianopsia or any obvious cognitive problems as evaluated with the Mini-Mental State examination
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital

Exclusion Criteria:

* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal disorders, or disorders from systematic diseases other than stroke

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-01; Study Completion 2007-12

PRIMARY OUTCOMES:
To investigate the balance recovery(proactive postural adujustments and reactive postural reaction) post-onset of each stroke subject

SECONDARY OUTCOMES:
To investigate the incidence of falls before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan Unversity Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan